CLINICAL TRIAL: NCT04719247
Title: Clinical and Radiographic Evaluation of Turmeric, Thymus Vulgaris, Nigella Sativa and Aloe Vera as Pulpotomy Medicaments in Primary Teeth" A Randomized Controlled Study
Brief Title: Clinical and Radiographic Evaluation of Turmeric, Thymus Vulgaris, Nigella Sativa and Aloe Vera as Pulpotomy Medicaments in Primary Teeth
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana sharaf, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PED19-3D
Record Dates: First submitted 2020-10-09; First posted 2021-01-22 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Turmeric (Experimental): Turmeric extract will be used as a dental pulp dressing material after pulpotomy and compared with Formocresol
  Interventions: Procedure: Pulpotomy
- Thymus Vulgaris (Experimental): Thymus Vulgaris extract will be used as a dental pulp dressing material after pulpotomy and compared with Formocresol
  Interventions: Procedure: Pulpotomy
- Nigella Sativa (Experimental): Nigella Sativa extract will be used as a dental pulp dressing material after pulpotomy and compared with Formocresol
  Interventions: Procedure: Pulpotomy
- Aloe Vera (Experimental): Aloe Vera extract will be used as a dental pulp dressing material after pulpotomy and compared with Formocresol
  Interventions: Procedure: Pulpotomy
- Formocresol (Active Comparator): Formocresol will be used as a dental pulp dressing material after pulpotomy to be compared with other materials.
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy — Irreversibly damaged dental pulp is partially removed and a dressing either Turmeric or Thymus Vulgaris or Nigella Sativa or Aloe Vera is placed. Clinical and Radiographic signs and symptoms are assessed and compared with Formocresol.

SUMMARY:
when caries reaches the pulp of the tooth, it has to be removed and replaced with a material. In this study im examining the clinical and radiographic signs and symptoms after using different natural materials in pulpotomized molars and compared to the formocresol.

DETAILED DESCRIPTION:
Patients who have irreversible pulpitis and need pulpotomy will be selected randomly from the out patient clinic. they will be assigned randomly to different study and control groups. pulpotomy will be performed in the second primary molar and 1 of the five materials will be put in the pulp chamber (aloe vera, nigella sativa, thymus vulgaris, turmeric and formocresol). It will be covered with a restoration and a stainless steel crown. Patients follow up will be done after 1,3,6 and 12 months to assess clinical and radiographic signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 4 to 7 years old
* Patients who are medically free
* Patients who have a restorable vital deep carious primary molar which is indicated for pulpotomy.
* No clinical signs or symptoms as pain on percussion, tooth mobility, presence of sinus or fistula, history of swelling.
* No radiographic signs of any periapical pathosis or signs of internal or external root resorption.

Exclusion Criteria:

* Patients who have any medical condition.
* Teeth that are badly broken down, that cannot be restored.
* Presence of uncontrolled bleeding.
* Clinical evidence of non-vitality such as presence of an abscess or a sinus or premature mobility.
* Radiographic evidence of bone resorption, internal or external root resorption and periapical or interradicular radiolucency.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical signs and symptoms of pulp reaction | 1 to 6 months
  Evaluated using Zurn and Seale criteria. (pain, infection, gingival health, tooth mobility) where 1 indicates asymptomatic and 4 indicates severe discomfort
Radiographic signs of pulp reaction | 1 to 6 months
  Evaluated using Zurn and Seale criteria. (radiolucency, bone resorption, internal or external resorption) where 1 indicates no radiographic changes while 4 indicates the presence of pathologic changes

CONTACTS AND LOCATIONS:
Overall Officials: Noha S Kabil, PHD, Study Director — Professor; Basma G Awad, PHD, Study Director — Lecturer
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saikiran KV, Kamatham R, Sahiti PS, Nuvvula S. Pulpotomy medicaments in primary teeth: A literature reviewof natural alternatives. SRM J Res Dent Sci 2018; 9:181-5.
- [Background] Kumar Praveen NH, Nayak Rashmi, Bhaskar Vipin K, Mopkar Pujan P Pulpotomy Medicaments: Continued Search for New Alternatives- A Review. 2014; OHDM - Vol. 13 - No. 4
- [Background] Al-Dlaigan YH. Pulpotomy Medicaments used in Deciduous Dentition: An Update. J Contemp Dent Pract. 2015 Jun 1;16(6):486-503. doi: 10.5005/jp-journals-10024-1711. PMID 26323453
- [Background] Salman BN, Vahabi S, Rad MM. Use of herbs and medicinal plants in dentistry: a review. Journal Dental School 2017; 35, No. 2: 58-64
- [Background] Subramanyam D, Somasundaram S. Clinical and Radiographic Outcome of Herbal Medicine Versus Standard Pulpotomy Medicaments in Primary Molars: A Systematic Review. Journal of Clinical and Diagnostic Research 2017 Oct; 11(10): ZE12-ZE16
- [Background] Kumar G, Jalaluddin M, Rout P, Mohanty R, Dileep CL. Emerging trends of herbal care in dentistry. J Clin Diagn Res. 2013 Aug;7(8):1827-9. doi: 10.7860/JCDR/2013/6339.3282. Epub 2013 Aug 1. PMID 24086929
- [Background] Kuwatada JS, Raja M, Sood P. Turmeric: A Boon to Oral Health. Int J Oral Care Res 2017;5(4):338-341.
- [Background] Srivastava R, Jyoti B, Pathak S, Wazir S, Shukla A, Sajid MdZ Aloe Vera: The Herbal Magic Wand. J Clin Den Res Edu 2014; 3 (8).
- [Background] Huth KC, Paschos E, Hajek-Al-Khatar N, Hollweck R, Crispin A, Hickel R, Folwaczny M. Effectiveness of 4 pulpotomy techniques--randomized controlled trial. J Dent Res. 2005 Dec;84(12):1144-8. doi: 10.1177/154405910508401210. PMID 16304444